CLINICAL TRIAL: NCT01040442
Title: The Effect of Plantar Vibration Stimuli on the Balance of Older Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal de Sao Carlos (Other)
Responsible Party: Fábio da Silva Wanderley, Fábio da Silva Wanderley
Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: fabio wanderley
Expanded Access: Available
Record Dates: First submitted 2009-12-28; First posted 2009-12-29 (Estimated); Last update posted 2009-12-29 (Estimated); Status verified 2009-08

CONDITIONS: Deficit Elderly Women With Body Balance
Keywords: Postural Balance; Aging; Accidental Falls; Vibration

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- vibration stimuli (Experimental)
  Interventions: Other: vibration stimuli

INTERVENTIONS:
Other: vibration stimuli — A single physical therapist performed the intervention using a Novafon SK2‡ vibratory stimulation device at a frequency of 100 Hz and sway amplitude of 2 mm. The participants of the experimental group received vibratory stimulation, applied slowly by sliding the head of the device over the entire plantar region for ten minutes for each foot at every session. During the intervention, the participants remained in the supine position on an examination table.

SUMMARY:
The objective of the present study was to identify the effect of direct vibration at a frequency of 100 Hz, applied to the plantar region, on the balance of women aged 60 years or older. The hypothesis is that the place improves body balance.

ELIGIBILITY:
Inclusion Criteria:

* women aged 60 or older, static balance deficit verified by the One-Leg Stance test with eyes open (OLSeo) (inability to maintain position for 30 seconds with eyes open, which is associated with the risk of falling17), independent gait without the use of walking aids.

Exclusion Criteria:

* individuals undergoing treatment to improve balance, inability to understand verbal commands, pathologies that affect balance and gait, use of medication that may affect balance, lower limb surgery in the past 12 months or participation in a physical activity program.

Ages: 60 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2008-03; Primary Completion 2008-08 (Actual); Study Completion 2009-08 (Actual)

REFERENCES:
- [Derived] Wanderley FS, Alburquerque-Sendin F, Parizotto NA, Rebelatto JR. Effect of plantar vibration stimuli on the balance of older women: a randomized controlled trial. Arch Phys Med Rehabil. 2011 Feb;92(2):199-206. doi: 10.1016/j.apmr.2010.10.014. PMID 21272715